CLINICAL TRIAL: NCT02167906
Title: Impact of Hand Osteoarthritis on Arterial Stiffness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 9356
Record Dates: First submitted 2014-06-17; First posted 2014-06-19 (Estimated); Last update posted 2022-12-14 (Actual); Status verified 2014-06

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- hand oa patients (Experimental): assess the carotid-femoral arterial stiffness determined by measuring the PWV
  Interventions: Other: arterial stiffness measurement
- without Hand OA patients (Active Comparator): assess the carotid-femoral arterial stiffness determined by measuring the PWV
  Interventions: Other: arterial stiffness measurement

INTERVENTIONS:
Other: arterial stiffness measurement

SUMMARY:
Patients affected by osteoarthritis (OA) have an increase overall mortality compared to the general population, mainly due to cardiovascular diseases. OA patients without cardiovascular risk have a 10 years cardiovascular events higher of around 15-30 %. Although the molecular mechanisms are still not well known, the structure and function of the vessel wall can be affected by several inflammatory and metabolic parameters during OA.These functional and structural changes of the arterial wall leads to arterial stiffness, measured by the pulse-wave velocity (PWV). PWV is the most widely used technique to assess arterial stiffness and has been shown to have predictive value for morbidity and mortality. In our study, we planned to compare arterial stiffness in OA patients with healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical hand OA defined according to the ACR (American College of Rheumatology) criteria.
* Patients with radiographic hand OA defined according to the Kellgren
* Lawrence criteria (≥ 2).
* Steady dose of statins for at least one month.
* Subject affiliated to a social security scheme
* Written informed consent

Exclusion Criteria:

* Rheumatoid arthritis, psoriatic arthritis or other inflammatory arthritis diseases.
* History of arterial hypertension treated and / or uncontrolled (SBP > 140 mmHg and DBP (diastolic blood pressure) > 90 mmHg)
* Diabetes (fasting blood glucose > 7 mmol/L)
* Obesity (BMI > 35 kg/m²)
* Chronic renal failure defined by a glomerular filtration rate <60 ml/min/1,73m ².
* Patient with uncontrolled cardiovascular disease or a personal history of cardiovascular events (myocardial infarction and angina, occlusive arterial disease, stroke)
* Pregnant or breastfeeding, or premenopausal and not taking an effective contraception

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-09-01 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2019-10-16 (Actual)

PRIMARY OUTCOMES:
carotid-femoral arterial stiffness | within the first 15 days after inclusion
  To assess the carotid-femoral arterial stiffness determined by measuring the PWV in patients with hand OA compared to healthy subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- UH Montpellier, Montpellier, France